CLINICAL TRIAL: NCT03475836
Title: Volatile Terpenes and Brain Function: Investigation of the Cognitive and Mood Effects of Mentha Spicata/Piperita Essential Oil With in Vitro Properties Relevant to Central Nervous System Function
Brief Title: Cognitive Effects of Mint Essential Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, David Kennedy, Professor, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SUB052_Forster_040216
Record Dates: First submitted 2018-02-13; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Cognitive Change; Affect
Keywords: Mentha; Mint; Essential oil; Cognition; Mood; Humans
MeSH Terms: interventions — peppermint oil

STUDY DESIGN:
Intervention Model Description: Randomised, placebo controlled, crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind. Treatments were prepared and coded by a third party researcher who had no further involvement with the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Vegetable oil
  Interventions: Dietary Supplement: Placebo
- High-dose mint essential oil (Active Comparator): 100 μL Mentha piperita essential oil (in vegetable oil)
  Interventions: Dietary Supplement: Mentha piperita
- Low-dose mint essential oil (Active Comparator): 50 μL Mentha piperita essential oil (in vegetable oil)
  Interventions: Dietary Supplement: Mentha piperita

INTERVENTIONS:
Dietary Supplement: Mentha piperita — Commercially available essential oil suspended in an off-the-shelf vegetable oil.
  Other Names: Peppermint
  Arms: High-dose mint essential oil; Low-dose mint essential oil
Dietary Supplement: Placebo — Inert placebo control in the form of vegetable oil. This matches the vegetable oil in the active intervention condition.
  Arms: Placebo

SUMMARY:
This study investigates the cognitive and mood effects of mint essential oils in a group of healthy, human adults. The investigational product will also be tested in vitro to ensure a number of biological mechanisms.

DETAILED DESCRIPTION:
The volatile components of essential oils (e.g. sage, lemon balm and rosemary)are found to exert a number of psychotropic effects and the monoterpenes in particular seem to be responsible for the cognitive and mood effects attributed to them.

The current study aims to investigate the cognitive and mood effects of mint essential oil in humans and to ensure the efficacy of the investigational product by conducting in vitro analysis on central nervous system receptor binding properties.

This will be achieved by analysing gamma-Aminobutyric acid A (GABAA), neuronal nicotinic and N-methyl-D-aspartate receptor (NMDA) glutamate receptor binding efficacy, acetylcholinesterase (AChE) inhibition, and gas chromatography-mass spectrometry (GC-MS) analysis will quantify % Limonene, % Carvone, % Menthone and % Menthol levels in the investigational treatment.

Cognitive and mood assessment will be via a randomised, placebo controlled, crossover design in 24, healthy adults aged between 18-35 yrs which will involve x1 training and x3 testing visits to the lab (placebo, 50 (micro Litre) μL and 100 μL Mentha piperita essential oil).

ELIGIBILITY:
Inclusion Criteria:

* 18-35 yrs
* Free from illicit drugs, alcohol, prescription medication (apart from contraception in the case of women) and herbal extracts/food supplements at each assessment.

Exclusion Criteria:

* Head injury, neurological disorder or neuro-developmental disorder
* English not 1st language (or not equivalent to a native English speaker)
* Relevant food allergies/intolerances or digestive problems
* Smokes tobacco
* Drinks excessive amounts of caffeine (more than 600mg day as assessed by a caffeine consumption questionnaire)
* Takes illicit social drugs
* Pregnant, seeking to become so, or breast feeding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2016-06-09 (Actual); Study Completion 2016-06-09 (Actual)

PRIMARY OUTCOMES:
Changes in cognition | 1, 3 and 6 hrs post-dose
  Changes in cognitive function as assessed by the following tasks: immediate and delayed word and picture recognition; name to face recall; 'Sternberg' Numeric Working Memory task; Corsi blocks; serial 3 subtractions; serial 7 subtractions; rapid visual information processing; peg and ball and choice reaction time. All tasks provide an outcome measure of accuracy, speed and error.

SECONDARY OUTCOMES:
Changes in mood | 1, 3 and 6 hrs post-dose
  Changes in mood assessed via the Speilberger State-Trait Anxiety Inventory (STAI) and Bond-Lader visual analogue mood scales. Scores on both measures are calculated at baseline and scores from subsequent completions are subtracted from this to produce change (change from baseline) scores. For both STAI and Bond-Lader these are numerical scores.
Neurotransmitter receptor binding efficacy | 0 hrs
  In Vitro analysis of investigational product for GABAA, neuronal nicotinic and NMDA glutamate receptor binding efficacy utilizing radioligand competition binding assays
Acetylcholinesterase inhibition | 0 hrs
  In Vitro analysis of investigational product for acetylcholinesterase inhibition as described in Okello, Coleman and Seal (2015)
Quantification of monoterpene levels | 0 hrs
  In Vitro analysis of investigational product for levels of % Limonene, % Carvone, % Menthone and % Menthol utilizing Gas chromatography-mass spectrometry. The method is described in Abuhamdah et al. (2015).

CONTACTS AND LOCATIONS:
Overall Officials: David O Kennedy, PhD, Principal Investigator — Northumbria University

IPD SHARING:
Plan to Share IPD: Undecided
No plan is currently available